CLINICAL TRIAL: NCT00148044
Title: Uremic Toxins of Patients With Acute Kidney Failure
Status: Completed | Type: Observational
Sponsor: University Hospital, Ghent (Other)
Other Study IDs: 2003/298
Record Dates: First submitted 2005-09-06; First posted 2005-09-07 (Estimated); Last update posted 2007-12-28 (Estimated); Status verified 2007-12

CONDITIONS: Kidney Failure, Acute
MeSH Terms: conditions — Acute Kidney Injury | interventions — Blood Specimen Collection

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Blood sampling for determination of uremic toxins

SUMMARY:
Determination of the concentration of uremic toxins of sepsis patients with or without acute kidney failure compared to the concentrations of uremic toxins of chronically uremic patients

DETAILED DESCRIPTION:
Determination of the concentration of uremic toxins of sepsis patients with or without acute kidney failure compared to the concentrations of uremic toxins of chronically uremic patients

ELIGIBILITY:
Inclusion Criteria:

* Intensive Care patients with sepsis
* Patients with acute kidney failure: serum creatinin > 2 mg/dl
* Chronic haemodialysis patients

Exclusion Criteria:

* < 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30
Dates: Start 2003-10; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Vanholder, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (1):
- University Hospital Ghent, Ghent, Belgium

REFERENCES:
- See also: Website University Hospital Ghent — http://www.uzgent.be